CLINICAL TRIAL: NCT05021601
Title: Bi-atrial Versus Left Atrial Ablation for Patients With Rheumatic Mitral Valve Disease and Non-paroxysmal Atrial Fibrillation: a Multicenter, Prospective, Randomized Controlled Trial
Brief Title: Bi-atrial Versus Left Atrial Ablation for Patients With Rheumatic Mitral Valve Disease and Non-paroxysmal Atrial Fibrillation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-1515
Record Dates: First submitted 2021-08-16; First posted 2021-08-25 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Persistent Atrial Fibrillation
Keywords: Rheumatic mitral valve disease; Surgical ablation; Mitral valve surgery
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bi-atrial ablation group (Experimental): Participants in this group will receive mitral valve surgery concomitant with bi-atrial ablation procedure.
  Interventions: Procedure: Bi-atrial ablation
- Left atrial ablation group (Active Comparator): Participants in this group will receive mitral valve surgery concomitant with left atrial ablation procedure.
  Interventions: Procedure: Left atrial ablation

INTERVENTIONS:
Procedure: Bi-atrial ablation — This intervention includes mitral valve surgery concomitant with left atrial ablation and right atrial ablation.
  Arms: Bi-atrial ablation group
Procedure: Left atrial ablation — This intervention includes mitral valve surgery concomitant with left atrial ablation alone.
  Arms: Left atrial ablation group

SUMMARY:
This study is aimed to compare the efficacy of bi-atrial ablation with left atrial ablation for atrial fibrillation during mitral valve surgery in patients with rheumatic mitral valve disease.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is present in 40%-60% of patients with rheumatic mitral valve disease (RMVD), which is an independent predictor of mortality and late stroke. During mitral valve (MV) surgery, the open left atrium facilitates a bi-atrial ablation procedure. However, a simplified lesion set including isolated pulmonary vein isolation or posterior left atrial (LA) wall isolation or LA maze was usually applied. The current literatures provide insufficient evidence to determine the potential benefits of bi-atrial ablation procedure when comparing with LA ablation procrdure in patients with non-paroxysmal AF and RMVD.

Patients with RMVD often have longer history, which tends to affect the right atrium, including pulmonary hypertension or tricuspid regurgitation.The necessity of bi-atrial ablation procedure targeting the bi-atrial substrate for AF in RMVD requires to be explored. In this study, we aimed to compare the efficacy of bi-atrial ablation with LA ablation for AF during MV surgery in patients with RMVD.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosis of persistent atrial fibrillation(AF) or long-standing persistent AF by medical history and Holter monitoring (persistent AF lasting more than 7 days; long-standing persistent AF lasting more than 1 year).
* Rheumatic mitral valve disease(RMVD) requires mitral valve surgery( RMVD was determined by history of acute rheumatic fever, valve morphology, echocardiographic findings and pathological diagnosis).
* Consent to surgical ablation of AF

Exclusion Criteria:

* Paroxysmal AF
* Degenerative or ischemic mitral valve disease
* Evidence of active infection
* Previous catheter ablation or surgical ablation for AF
* Surgical management of hypertrophic obstructive cardiomyopathy
* Absolute contraindications for anticoagulation therapy
* Left atrial thrombosis (not including left atrial appendage thrombosis alone)
* Chronic obstructive pulmonary disease(Forced expiratory volume in 1 second (FEV1)<30% anticipated value)
* Uncontrolled hypo- or hyperthyroidism
* Mental impairment or other conditions that may not allow participants to understand the nature, significance, and scope of study
* Left atrial diameter>70mm
* Right ventricular dysfunction (TAPSE<16) or moderate to severe tricuspid regurgitation or pulmonary artery pressure (estimated by echocardiography) >60mmHg
* Coronary artery bypass grafting is required for participants with coronary heart disease
* Previous cardiac surgery
* Refuse to participate in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2022-05-10 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Survival rate without any recurrence of atrial tachyarrhythmias in the absence of antiarrhythmic drugs | At 12-month after intervention
  Without detections of atrial fibrillation, atrial flutter, or other atrial tachyarrhythmias with a duration of greater than 30 seconds documented by 3-day Holter monitoring in the absence of antiarrhythmic drugs.

SECONDARY OUTCOMES:
Survival rate without permanent pacemaker implantation (Key secondary outcome) | At 12-month after intervention
  Percentage of participants who did not have a new permanent pacemaker implanted.
Survival rate without any recurrence of atrial tachyarrhythmias with antiarrhythmic drugs | At 12-month after intervention
  Without detections of atrial fibrillation, atrial flutter, or other atrial tachyarrhythmias with a duration of greater than 30 seconds documented by 3-day Holter monitoring with antiarrhythmic drugs.
Burden of atrial fibrillation | At 12-month after intervention
  Burden of atrial fibrillation according to 3-day Holter monitoring.
Major adverse events | At 12-month after intervention
  Including cardiac death, stroke, heart failure requiring rehospitalization, embolic events or bleeding events requiring rehospitalization.
Cardiac function | At 12-month after intervention
  Documented by echocardiography (left ventricular ejection fraction).

CONTACTS AND LOCATIONS:
Overall Officials: Zhe Zheng, MD,PhD, Study Chair — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (2):
- China (2):
  - Fuwai Hospital, Beijing, Beijing Municipality
  - Nanjing First Hospital, Nanjing Medical University, Nanjing, Jiangsu

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yu C, Li H, Wang Y, Chen S, Zhao Y, Zheng Z. Bi-atrial versus left atrial ablation for patients with rheumatic mitral valve disease and non-paroxysmal atrial fibrillation (ABLATION): rationale, design and study protocol for a multicentre randomised controlled trial. BMJ Open. 2022 Nov 29;12(11):e064861. doi: 10.1136/bmjopen-2022-064861. PMID 36446460